CLINICAL TRIAL: NCT04502615
Title: Effect of Sand on Knee Load and sEMG Activity During a Single Leg Landing Task: Implications for ACL Prevention and Rehabilitation
Brief Title: Effect of Sand on Knee Load and Muscle Activity During a Single Leg Landing Task
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Responsible Party: Principal Investigator, Mark Richardson, Principal Investigator, Teesside University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TeessideUni
Record Dates: First submitted 2020-07-30; First posted 2020-08-06 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Single Leg Hop Sand Surface; Single Leg Hop Grass Surface; Single Leg Hop Firm Surface
Keywords: Sand; knee valgus; knee abduction moment; electromyography
MeSH Terms: interventions — Sand

STUDY DESIGN:
Intervention Model Description: Randomised, repeated measures crossover design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sand (Experimental): Participants perform 5 single leg hops onto a Sand surface from a 30cm height
  Interventions: Other: Sand
- Artificial grass (Active Comparator): Participants perform 5 single leg hops onto a grass surface from a 30cm height
  Interventions: Other: artificial grass
- Firm Ground (Active Comparator): Participants perform 5 single leg hops onto a firm ground surface from a 30cm height
  Interventions: Other: firm ground

INTERVENTIONS:
Other: Sand — sand surface
  Arms: Sand
Other: artificial grass — grass surface
  Arms: Artificial grass
Other: firm ground — firm surface
  Arms: Firm Ground

SUMMARY:
This study evaluates the effect of different surfaces on the load experienced by the knee when landing from a single leg hop. A sand, pliable grass and firm (hard floor) surface will be compared when hopping from a 30 cm height. Each subject will complete 5 hops on each surface in a random order. The muscle activity in selected muscles of the lower limb will also be investigated to see how this differs in the landing leg, when landing on the different surfaces.

DETAILED DESCRIPTION:
The aim of this study is twofold: 1) To investigate the effect of sand on landing kinematics and kinetics at the knee joint when performing a single leg jump landing task (dominant leg), comparing sand with a firm surface and pliable grass control. 2) To investigate the sEMG activity of the hamstring, quadriceps and gastrocnemius muscles of the dominant leg during the jump landing task on these different surfaces (from take off through to terminal knee flexion at the end of the landing phase).

ELIGIBILITY:
Inclusion Criteria:

* Female
* Participate in a minimum of 3 hours sporting activity per week.
* Provided Informed Consent
* Must be over 16 years of age (16-45 years)
* No exclusion criteria

Exclusion Criteria:

* Not willing to provide informed consent
* Pregnant
* History of ACL injury or other knee pathology
* Significant lower limb pathology
* Previous lower limb fracture or surgery
* Lower Limb injury in last 3 months.
* Male

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — most be female to be eligible for the study
Enrollment: 20 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
knee abduction moment (N.m) | 1 testing session (1 day)
  a combination of ground force and amount of knee valgus on landing
knee valgus | 1 testing session (1 day)
  angle at the knee on landing
surface electromyography (sEMG) activity pre and post landing | 1 testing session (1 day)
  muscle activity of quadriceps (vastus medialis, vastus lateralis), hamstrings (lateral and medial), gastroc (lateral head)

SECONDARY OUTCOMES:
Anterior tibial translation | 1 testing session(1 day)
  The amount of forward translation of the tibia when landing on the surface

CONTACTS AND LOCATIONS:
Overall Officials: Mark Richardson, MSc, Principal Investigator — Teesside University
Locations (1):
- Teesside University, Middlesbrough, United Kingdom

REFERENCES:
- [Derived] Richardson MC, Evans W, Chesterton P, Wright M. The effects of a 6-week sand- vs. Land-based jump training programme on frontal plane knee angle and jump performance in adolescent female football players. J Sports Sci. 2025 Mar;43(6):523-535. doi: 10.1080/02640414.2025.2465946. Epub 2025 Feb 18. PMID 39964088